CLINICAL TRIAL: NCT05646030
Title: Feasibility, Reliability, and Satisfaction of Carcinoembryonic Antigen Measurements Using Home Based (automated) CApillary Blood SAmpling; the Prospective CASA-I Study
Brief Title: Feasibility, Reliability, and Satisfaction of CEA Using Home Based (automated) Capillary Blood Sampling
Acronym: CASA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, D.J. (Dirk) Grünhagen, Principal Investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NL78309.078.21
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: Capillary sampling; CEA; Colorectal cancer; Home-based
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Phlebotomy

STUDY DESIGN:
Intervention Model Description: A prospective three-armed cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Subjects with known elevated serum CEA (Other): Before the start of sample collection questionnaire A on paper will be filled in by all study subjects. The order of sample collection will be: automated capillary sampling, lancet capillary sampling and venipuncture. Herein automated and lancet capillary sampling will be performed by the study subjects themselves whereas the venipuncture will be performed by the study personnel. After all sampling has been completed, the subject is asked to complete questionnaire B which will evaluate pain, burden, ease of use and preference.
  For subjects in arm A and C this entails the end of the study
  Interventions: Diagnostic Test: TAP-II; Diagnostic Test: Lancet capillary sampling; Diagnostic Test: Venipuncture
- Subjects currently undergoing colorectal cancer related follow-up (Other): The subjects of arm B are requested to perform automated capillary and lancet capillary sampling at home following their next two outpatient visits. During these outpatient visits, a reference value blood CEA measurement will be obtained using venipuncture by the personnel of the clinical laboratory of Erasmus MC. The required materials will be sent to the home address of the patient. Sampling will be performed at home and by the subjects themselves. Subjects will have access to the tutorial videos for automated and lancet capillary sampling.
  Interventions: Diagnostic Test: TAP-II; Diagnostic Test: Lancet capillary sampling; Diagnostic Test: Venipuncture
- Volunteers (Other): Before the start of sample collection questionnaire A on paper will be filled in by all study subjects. The order of sample collection will be: automated capillary sampling, lancet capillary sampling and venipuncture. Herein automated and lancet capillary sampling will be performed by the study subjects themselves whereas the venipuncture will be performed by the study personnel. After all sampling has been completed, the subject is asked to complete questionnaire B which will evaluate pain, burden, ease of use and preference.
  For subjects in arm A and C this entails the end of the study
  Interventions: Diagnostic Test: TAP-II; Diagnostic Test: Lancet capillary sampling; Diagnostic Test: Venipuncture

INTERVENTIONS:
Diagnostic Test: TAP-II — The TAP-II device will be compared to lancet capillary sampling and the venipuncture
Diagnostic Test: Lancet capillary sampling — The lancet capillary sampling will be compared to TAP device and the venipuncture
Diagnostic Test: Venipuncture — The venipuncture will be compared to TAP device and the lancet capillary sampling

SUMMARY:
The goal of this study is to determine the feasibility of CEA assessments at home using (automated) capillary sampling in patients in the follow-up after treatment for colorectal cancer.

The main questions it aims to answer are:

* To determine the success rate of capillary sampling at home by the patient
* To assess reliability and satisfaction of (automated) capillary CEA measurements Participants will be asked to perform automated capillary sampling and lancet capillary sampling at home twice after regular check-up visits in the hospital, with an interval of 3-6 months in between. During this hospital visit, a CEA measurement in blood sampled by venipuncture will be performed to act as a reference for the CEA measurements in (automated) capillary blood to be sampled at home.

Reliability of CEA measurements will be assessed for automated capillary and lancet capillary sampling compared to venipuncture.

Satisfaction in terms of patient reported outcomes (pain, burden, ease of use, and preference) will be evaluated.

DETAILED DESCRIPTION:
The follow-up of patients after colorectal cancer surgery mainly consists of blood CEA assessments. These blood assessments could be done at home and could be beneficial in terms of patients' well-being and societal cost-effectiveness. Capillary blood sampling can be an alternative to venipuncture in home based or decentralized surveillance as it can be performed by the patient themselves. Before home based capillary sampling can be implemented, feasibility, reliability, and satisfaction for serum CEA measurements has to be determined.

ELIGIBILITY:
Inclusion Criteria:

Arm A: subjects with known elevated serum CEA

* Age ≥ 21 years
* Histologically confirmed (metastatic) colorectal adenocarcinoma
* Serum CEA ≥ 10 μg/L within the last 2 months determined using venipuncture blood sampling

Arm B: subjects currently undergoing colorectal cancer related follow-up

* Age ≥ 21 years
* Histologically confirmed (metastatic) colorectal adenocarcinoma
* Currently undergoing in-hospital follow-up with at least two more scheduled serum CEA assessments 3-6 months apart

Arm C: volunteers

* Age ≥ 21 years
* No known history of colorectal adenocarcinoma
* No known history of elevated serum CEA ≥ 5 μg/L

Exclusion Criteria:

* Illiteracy and/or insufficient proficiency of the Dutch language
* Severe or complete loss of sensory and or motor function of one or both arms and or hands
* Known medical history of superficial or deep skin infection after venipuncture or intravenous line that required antibiotic treatment and or hospital admittance
* Known medical history of immunodeficiency or current use of medical immunosuppressants
* Known medical history of blood-borne diseases such as but not limited to the human immunodeficiency virus, hepatitis and viral hemorrhagic fever

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of CEA assessments at home using (automated) capillary sampling | Year 1 (6 months after the inclusion of the first patient)
  Home based (automated) capillary sampling will be considered feasible if a success rate of 85% or greater has been reached. Herein a successful (automated) capillary sampling at home is defined as a sampling of blood by the patient that reached the clinical laboratory of the hospital via post and in which a CEA level could be determined reliably. Both capillary sampling methods will be analysed and compared to venepuncture separately.

SECONDARY OUTCOMES:
Reliability of the CEA measurements | Year 1 (6 months after the inclusion of the first patient)
  Reliability will be assessed by a Bland-Altman analysis to determine mean bias and the 95% limits of agreement of measurements from (automated) capillary samples compared to venipuncture samples. These will be compared to predefined clinically relevant cut-off values for the mean bias and the limits of agreement. A mean bias of greater or equal to +/- 5% and or 95% limits of agreement equal to or greater than +/- 10% will be considered clinically relevant and thereby unreliable. These cut-off values are defined based on previously found 95% limits of agreement of the automated capillary sampling device and the precision of the Cobas 8000 analyzer which will be used to perform the CEA analyses.
Satisfaction of blood sampling | Year 1 (6 months after the inclusion of the first patient)
  All study subjects will be asked to complete the questionnaire to evaluate pain, burden, ease of use and preference. Herein they are asked to provide their perceived level of pain separately for automated capillary sampling, lancet capillary sampling and venipuncture. A visual analogue scale ranging from 0 to 10 will be used to measure perceived level of pain. Pain measurements will be compared across all three sampling methods in the entire cohort of 100 subjects using repeated measures ANOVA. An α < 0.05 will be considered statistically significant.
Clinical laboratory sample processing time: | Year 1 (6 months after the inclusion of the first patient)
  the sample processing time from entering the clinical laboratory until a successful measurement is obtained will be compared across all sampling methods using analysis of variance (ANOVA). An α < 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Grünhagen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voigt KR, Wullaert L, Verhoef C, Grunhagen DJ, Ramakers C. Reliable capillary sampling of carcinoembryonic antigen at home: the CASA feasibility study. Colorectal Dis. 2023 Jun;25(6):1163-1168. doi: 10.1111/codi.16536. Epub 2023 Mar 21. PMID 36945082
- [Background] Voigt KR, Wullaert L, Gobardhan PD, Doornebosch PG, Verhoef C, Husson O, Ramakers C, Grunhagen DJ. Feasibility, reliability and satisfaction of (automated) capillary carcinoembryonic antigen measurements for future home-based blood sampling: the prospective CASA-I study. Colorectal Dis. 2024 Aug;26(8):1560-1568. doi: 10.1111/codi.17085. Epub 2024 Jul 1. PMID 38949106